CLINICAL TRIAL: NCT06189651
Title: Short-Term Efficacy of 5% Dextrose Injection With Ultrasound Guided Nerve Hydrodissection Method in Carpal Tunnel Syndrome: Prospective Randomized Controlled Study
Brief Title: Short Term Efficacy of 5% Dextrose Injection With Ultrasound Guided Nerve Hydrodissection Method in CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nazlı Derya Bugdayci, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STEDIUGNHMCTS
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; hydrodissection; 5% dextrose; wrist splint
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, clinical trials
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wrist splint treatment (Experimental): The same type of wrist splint was given
  Interventions: Device: wrist splint
- Wrist splint treatment+ %5 dextrose injection (Experimental): The same type of wrist splint was given and 5% dextrose injection using USG-guided nerve hydrodissection method was applied
  Interventions: Device: wrist splint; Procedure: 5% dextrose injection using USG-guided nerve hydrodissection method

INTERVENTIONS:
Device: wrist splint — The same type of wrist splint to be used for at least 8 hours at night for 4 weeks, to be worn in a neutral position and in accordance with the wrist as described in previous studies to restrict movement in the wrist. Patients who did not sleep for 8 hours were asked to complete 8 hours of wrist splint use before going to sleep or after waking up.
Procedure: 5% dextrose injection using USG-guided nerve hydrodissection method — 2 ml each of 5% dextrose injection was administered once at the proximal wrist level above the median nerve separating the median nerve from the flexor retinaculum and below the median nerve separating the median nerve from the flexor tendons by nerve hydrodissection method in the transverse inplane plane under ultrasound guidance. After the application, the spread of the injectate was observed by looking longitudinally at the median nerve.
  Arms: Wrist splint treatment+ %5 dextrose injection

SUMMARY:
Hydrodissection injection method; It is a safe and effective injection method in peripheral nerve compression that aims to release the adhesions by separating the nerve from the surrounding connective tissues through the liquid given by injection. Perineural injection of 5% dextrose is analgesic in neuropathic pain, although the mechanism is not fully defined. USG-guided 5% dextrose injection using nerve hydrodissection method is promising in the treatment of CTS. In our study, we aimed to investigate the short-term (4 weeks) efficacy of 5% dextrose injection using USG-guided nerve hydrodissection method in combination with wrist splint treatment in patients with mild to moderate carpal tunnel syndrome (CTS) and whether this treatment can provide additional benefit to wrist splint treatment.

DETAILED DESCRIPTION:
In our prospective randomized controlled study, 44 patients who met the inclusion criteria and had mild to moderate carpal measured syndrome with EMG as described in previous studies were included in the study. The 44 volunteer participants with mild to moderate carpal tunnel syndrome were randomly divided into 2 groups as wrist splint treatment group (control group) and wrist splint + 5% dextrose injection treatment group (study group) by stratified and block randomization method. Stratified randomization was done according to the variable of having mild and moderate carpal tunnel syndrome. Assignment to the treatment or control group for each stratum was done by 1:1 block randomization.

All patients were given the same type of wrist splint to be used for at least 8 hours at night for 4 weeks, to be worn in a neutral position and in accordance with the wrist as described in previous studies to restrict movement in the wrist, and activities that aggravate symptoms (repetitive and demanding wrist movements: Knitting, keyboard use, use of vibrating tools, etc.) were recommended to be avoided. The given wrist splint is a commercially available wrist splint with a metal bar on the palmar side and Velcro straps on the dorsal side that can be adjusted according to the wrist, restricting flexion and extension of the wrist and allowing movement of the metacarpophalangeal joint. Patients who did not sleep for 8 hours were asked to complete 8 hours of wrist splint use before going to sleep or after waking up. All patients were given a wrist splint diary and asked to write down the days and hours of splinting. Patients who did not wear splints for enough days and hours were excluded from the study. In the study group, 2 ml each of 5% dextrose injection was administered once at the proximal wrist level above the median nerve separating the median nerve from the flexor retinaculum and below the median nerve separating the median nerve from the flexor tendons by nerve hydrodissection method in the transverse inplane plane under ultrasound guidance. After the application, the spread of the injectate was observed by looking longitudinally at the median nerve. A 25 gauge syringe was used for administration. Patients were observed for side effects and side effects were noted. Patients were asked to rate their injection pain on a Visual Analog Scale (VAS) after injection to measure the pain during injection. All patients were advised not to take any additional treatment for their symptoms during the study. Patients who received additional treatment were noted. All patients were evaluated with Visual Analog Scale (VAS) score, Turkish version of Boston Carpal Tunnel Questionnaire (BCTQ), grip strength (GS) measured by hand dynamometer, and median nerve cross-sectional area (CSA) measured by ultrasonography before the start of the study (week 0) and at the end of the 4th week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms for at least 3 months
* Patients with paresthesia or dysesthesia in the fingers
* Patients diagnosed with mild or moderate carpal tunnel syndrome by EMG

Exclusion Criteria:

* Patients with severe carpal tunnel syndrome
* Patients with polyneuropathy, cervical radiculopathy, brachial plexopathy and thoracic outlet syndrome
* Patients with a history of wrist surgery
* Patients within 6 months of steroid injection for carpal tunnel syndrome
* Patients with infection at the treatment site
* Patients with coagulation disorders or on coumadin
* Pregnant patients
* Patients with a history of malignancy, rheumatologic disease
* Patients with any other painful pathology in the upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Start of the study (week 0) and at the end of the 4th week.
  VAS was used to measure the severity of pain-paresthesia. Patients were given a white paper with a horizontal straight line with numbers from 0 to 10. The patients were told that the left-hand side of the line described gradually decreasing pain and the right-hand side described gradually increasing pain and that a score of 0 corresponded to no pain-paresthesia and a score of 10 corresponded to intolerable pain-paresthesia and were asked to mark a number on the scale.
Boston Carpal Tunnel Questionnaire (BCTQ) | Start of the study (week 0) and at the end of the 4th week.
  The BCTQ includes an eleven-question symptom severity scale (BCTQS) and an eight-question functional status scale (BCTQF) that assesses the degree of difficulty in daily activities. Symptom severity ranges from 11 (no symptoms) to 55 (severe symptoms). The functional status scale ranges from 8 (least difficulty) to 40 (maximum difficulty). Turkish version has been tested for reliability and validity.

SECONDARY OUTCOMES:
Grip Strength (GS) | Start of the study (week 0) and at the end of the 4th week.
  Maximal voluntary grip strength (GS) was measured with a hand dynamometer. This measurement was performed as described in previous studies; sitting, shoulders in adduction and neutral position, elbow in 90° flexion, forearm and wrist in neutral position. The measurements were performed three times. For each measurement, patients were asked to perform a maximal voluntary grip for five seconds. A rest period of 10 seconds was given between the three tests. The measurements were performed with a JAMAR Plus+ (by Sammons Preston) hand dynamometer. The average of these three measurements was used in the analysis. Before the test measurements, the patient was shown how to use the device practically.
Median Nerve Cross Sectional Area (CSA) | Start of the study (week 0) and at the end of the 4th week.
  CSA was measured axially on the wrist at the scaphoid-psiform bone level. The measurement results were expressed in mm2. CSA measurements were performed by the same investigator. In order to determine the level of intra-observer error, CSA measurements were performed twice in 10 subjects with an interval of one day. Intraobserver error was calculated using the technical error of measurements (TEM) method.

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Derya Bugdayci, Assoc. Prof., Study Director — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)